CLINICAL TRIAL: NCT03596177
Title: An Exploratory Phase 2a, Randomised, Double-blind, Placebo-controlled Study to Evaluate the Effect of MEDI0382 on Energy Balance in Overweight and Obese Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Effect of MEDI0382 on Energy Balance in Overweight and Obese Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5670C00021
Record Dates: First submitted 2018-06-11; First posted 2018-07-23 (Actual); Results first posted 2021-01-15 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-12

CONDITIONS: Diabetes Mellitus, Type II; Obesity
Keywords: Diabetes Mellitus, Type II; Obesity; MEDI0382
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — cotadutide

STUDY DESIGN:
Intervention Model Description: Randomised, Double-Blind, Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MEDI0382 (Experimental): Participants will receive subcutaneous (SC) injection of placebo for 16 days in the single-blind treatment period, and then SC injection of MEDI0382 titrated up to 300 μg for 42 days (100 μg for 4 days, followed by 200 μg for 4 days, and finally 300 μg for 34 days) in double-blind treatment period.
  Interventions: Drug: MEDI0382; Drug: Placebo
- Placebo (Placebo Comparator): Participants will receive SC injection of placebo for 16 days in the single-blind treatment period, and then SC injection of placebo matched to MEDI0382 for 42 days in double-blind treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MEDI0382 — MEDI0382 will be administered subcutaneously, titrated up to 300 μg for 42 days (100 μg for 4 days, followed by 200 μg for 4 days, and finally 300 μg for 34 days) in double-blind treatment period.
  Arms: MEDI0382
Drug: Placebo — Placebo will be administered subcutaneously for 16 days in the single-blind treatment period in both MEDI0382 and placebo arms, and SC injection of placebo matched to MEDI0382 for 42 days in double-blind treatment period in placebo arm.

SUMMARY:
An exploratory study to evaluate the effect of MEDI0382 on energy balance in overweight and obese participants with type 2 diabetes mellitus

DETAILED DESCRIPTION:
An exploratory Phase 2a, randomised, double-blind, placebo-controlled study to evaluate the effect of MEDI0382 on energy balance in overweight and obese participants with type 2 diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged >= 30 and <= 75 years at screening
2. Provision of signed and dated written informed consent (except for consent for genetic and non-genetic research and additional optional assessments) prior to any protocol-related procedures
3. Body Mass Index > 28 and <= 40 kg/m^2 at screening
4. Glycated haemoglobin (HbA1c) <= 8.0% at screening
5. Diagnosed with type 2 diabetes (T2DM) with glucose control managed with metformin, with or without a dipeptidyl peptidase 4 (DPPIV) inhibitor, Sodium-glucose co-transporter-2 inhibitors (SGLT2i), sulfonylurea, or meglitinide, where no significant dose change (increase or decrease > 50%) has occurred in the 3 months prior to screening; if the participant is on dual therapy, a 4-week washout of the non-metformin therapy (DPPIV inhibitor, SGLT2i, sulfonylurea, or meglitinide) will be required prior to Visit 4.
6. Female participants of childbearing potential must have a negative pregnancy test at screening and randomisation, and must not be lactating.
7. Female participants of childbearing potential who are sexually active with a non-sterilised male partner must be using at least one highly effective method of contraception from screening and must agree to continue using such precautions up until 4 weeks after the last dose of study drug

Exclusion Criteria:

1. History of, or any existing condition(s) that, in the opinion of the investigator, would interfere with evaluation of the study drug, put the participant at risk, influence the participant's ability to participate or affect the interpretation of the results of the study and/or any participant unable or unwilling to follow study procedures
2. Any participant with a cardiac pacemaker or implanted/portable electronic device
3. Any participant who has received another study drug as part of a clinical study or a Glucagon-like peptide-1 (GLP-1) analogue-containing preparation within the last 30 days or 5 half-lives of the drug (whichever is longer) at the time of screening (Visit 1)
4. Any participant who has received any of the following medications within the specified timeframe prior to Visit 2: herbal preparations or drugs licensed for control of body weight or appetite (eg, orlistat, bupropion, naltrexone, phentermine-topiramate, phentermine, lorcaserin, opiates, domperidone, metoclopramide, or other drugs known to alter gastric emptying)
5. Concurrent participation in another study with a study drug and prior randomisation in this study is prohibited
6. Severe allergy/hypersensitivity to any of the proposed study treatments, excipients, or standardised meals
7. Symptoms of acutely decompensated blood glucose control (eg, thirst, polyuria, weight loss), a history of type 1 diabetes mellitus or diabetic ketoacidosis, or if the participant has been treated with daily SC insulin within 90 days prior to screening.
8. Abnormal thyroid stimulating hormone (TSH) level of < 0.03 Milli-International Units Per Litre (mIU/L) or > 10 mIU/L confirmed on two consecutive tests
9. Regularly engage in high intensity exercise at least three times per week or have done so in the prior three months
10. Clinically significant inflammatory bowel disease, gastroparesis or other severe disease or surgery affecting the upper gastrointestinal tract (including weight-reducing surgery and procedures) which may affect gastric emptying or could affect the interpretation of safety and tolerability data
11. Acute or chronic pancreatitis
12. Significant hepatic disease (except for nonalcoholic steatohepatitis or nonalcoholic fatty liver disease without portal hypertension or cirrhosis) and/or participants with any of the following results at screening:

    1. Aspartate transaminase (AST) >= 3 × upper limit of normal (ULN)
    2. Alanine transaminase (ALT) >= 3 × ULN
    3. Total bilirubin >= 2 × ULN
13. Impaired renal function defined as estimated glomerular filtration rate (eGFR) < 45 mL/minute/1.73 m^2 at screening (GFR estimated according to the Chronic Kidney Disease-Epidemiology Collaboration (CKD-EPI) or the Modification of Diet in Renal Disease (MDRD) using MDRD Study Equation isotope dilution mass spectrometry-traceable [International System of Units (SI) units]
14. Poorly controlled hypertension defined as:

    1. Systolic blood pressure (BP) > 180 mm Hg
    2. Diastolic BP or > 100 mm Hg After 10 minutes of supine rest and confirmed by repeated measurement at screening.

    Participants who fail BP screening criteria may be considered for 24-hour ambulatory BP monitoring at the discretion of the investigator. Participants who maintain a mean 24-hour BP <= 180/100 mmHg with a preserved nocturnal dip of > 15% will be considered eligible
15. Unstable angina pectoris, myocardial infarction, transient ischemic attack or stroke within 3 months prior to screening, or participants who have undergone percutaneous coronary intervention or a coronary artery bypass graft within the past 6 months or who are due to undergo these procedures at the time of screening
16. Severe congestive heart failure (New York Heart Association Class III or IV)
17. Basal calcitonin level > 50 ng/L at screening or history/family history of medullary thyroid carcinoma or multiple endocrine neoplasia
18. History of neoplastic disease within 5 years prior to screening, except for adequately treated basal cell, squamous cell skin cancer, or in situ cervical cancer
19. Any positive results for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV) antibody
20. Substance dependence or history of alcohol abuse and/or excess alcohol intake
21. Involvement of any AstraZeneca, Medimmune Ltd, contract research organization (CRO), or National Institute for Health Research/Wellcome Trust Cambridge Clinical Research Facility employee or their close relatives

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2019-12-22 (Actual); Study Completion 2019-12-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Cambridge, United Kingdom

REFERENCES:
- See also: D5670C00021 CSP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5670C00021&attachmentIdentifier=bf8d7d39-e3d7-4035-a973-30f83c2db923&fileName=D5670C00021-clinical-protocol-amendment-5-Redacted1.pdf&versionIdentifier=
- See also: D5670C00021 SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5670C00021&attachmentIdentifier=0fba087b-4c08-4dd3-a44f-0946d4df5d91&fileName=D5670C00021_Statistical_Analysis_Plan_Redacted_V2.0.pdf&versionIdentifier=
- See also: CSR Addendum synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5670C00021&attachmentIdentifier=e435c4b6-40df-49c5-9623-000e54c22d01&fileName=D5670C00021_CSR_Addendum_synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to COVID-19 pandemic a full analysis could not be performed due to logistical challenges and equipment failure and no further conclusions can be drawn. The results from the secondary analyses presented in this CSR Addendum do not impact any of the conclusions presented in the CSR, (Data cut off [DCO] 31 January 2020), see details in "Limitations and Caveats" section
Groups:
- Placebo: Participants received subcutaneous (SC) injection of placebo for 16 days in the single-blind treatment period, and then SC injection of placebo matched to MEDI0382 for 42 days in double-blind treatment period.
- MEDI0382: Participants received SC injection of placebo for 16 days in the single-blind treatment period, and then SC injection of MEDI0382 titrated up to 300 μg for 42 days (100 μg for 4 days, followed by 200 μg for 4 days, and finally 300 μg for 34 days) in double-blind treatment period.
Period: Single Blind Period
Arm/Group | Placebo | MEDI0382
Started | 9 | 19
Completed | 7 | 18
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other | 1 | 0
Period: Double Blind Period
Arm/Group | Placebo | MEDI0382
Started | 7 | 18
Completed | 7 | 12
Not Completed | 0 | 6
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other | 0 | 4
Not completed — Death during safety follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: As-treated population included all participants who received any dose of study drug and analyzed according to the treatment they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MEDI0382 | Total
Number analyzed (Participants) | 9 | 19 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.2 (7.2) | 59.5 (8.4) | 60.4 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 7 | 18 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 18 | 27
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 0 | 1
  White | 8 | 18 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Body Weight From Baseline to Day 59
Description: Percent change in body weight from baseline to Day 59 is reported. Day 17 was considered as baseline for this outcome measure. The last observation carried forward (LOCF) analysis was used for missing data imputation for Day 59.
Time Frame: Baseline (Day 17) and Day 59
Population: Modified intent-to-treat (ITT) population: Participants in ITT population (who received any study drug) who received at least one dose of the study drug in the double-blind treatment period, and analyzed according to their randomized treatment group. Here, "number of participants analyzed" denotes those participants who were evaluable at baseline and Day 59.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent change in body weight
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 7 | 14
Percent change in body weight | -1.40 [-2.66 to -0.13] | -3.98 [-4.85 to -3.10]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382; Test type: Superiority; p = 0.011, ANCOVA; Mean Difference (Net) = -2.58, 90% CI 2-sided [-4.15 to -1.00]

2. Secondary Outcome: Percent Change in Total Energy Intake From the ad Libitum Lunch From Baseline to Day 32 and Day 59
Description: Total energy intake in kilojoules (kJ) were recorded in a food diary after ad libitum lunch on Days 16, 32, and 59. The ad libitum lunch was a standardised solid meal with food of known macronutrient content. Participants were advised to eat freely until they feel comfortably full and the meal duration was flexible according to participant's preference. During the meal, the quantity of food ingested was recorded by study site staff without participants' awareness that food consumption was recorded. Percent change in total energy intake from the ad libitum lunch is reported. Day 16 was considered as baseline for this outcome measure. The LOCF analysis was used for missing data imputation for Day 59.
Time Frame: Baseline (Day 16), Day 32, and Day 59
Population: mITT population: Participants in the ITT population (who received any study drug) who received at least one dose of the study drug in the double-blind treatment period, and analyzed according to their randomized treatment group. Here, "number of participants analyzed" denotes those participants who were evaluable at baseline and Days 32 and 59.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent change in total energy intake
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 7 | 14
Percent change in total energy intake
  Percent change at Day 32 | -5.170 [-23.344 to 13.003] | -50.652 [-63.480 to -37.823]
  Percent change at Day 59 | -10.598 [-31.316 to 10.119] | -51.922 [-66.546 to -37.297]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382; Statistical Analysis for Day 32; Test type: Superiority; p = 0.002, ANCOVA; Mean Difference (Net) = -45.481, 90% CI 2-sided [-67.777 to -23.186]
Statistical Analysis 2: Comparison: Placebo vs MEDI0382; Statistical Analysis for Day 59; Test type: Superiority; p = 0.011, ANCOVA; Mean Difference (Net) = -41.323, 90% CI 2-sided [-66.740 to -15.907]

3. Secondary Outcome: Change in Total Energy Intake From the ad Libitum Lunch From Baseline to Day 32 and Day 59
Description: Total energy intake in kilojoules (kJ) were recorded in a food diary after ad libitum lunch on Days 16, 32, and 59. The ad libitum lunch was a standardised solid meal with food of known macronutrient content. Participants were advised to eat freely until they feel comfortably full and the meal duration was flexible according to participant's preference. During the meal, the quantity of food ingested was recorded by study site staff without participants' awareness that food consumption was recorded. Change in total energy intake from the ad libitum lunch is reported. Day 16 was considered as baseline for this outcome measure. The LOCF analysis was used for missing data imputation for Day 59.
Time Frame: Baseline (Day 16) to Day 32 and Day 59
Population: as for outcome 2
Measure: Least Squares Mean (90% Confidence Interval); unit: Kilojoules
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 7 | 14
Kilojoules
  Change at Day 32 | -126.271 [-647.387 to 394.846] | -1677.465 [-2045.322 to -1309.607]
  Change at Day 59 | -410.816 [-1107.896 to 286.263] | -1743.331 [-2235.400 to -1251.261]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382; Statistical Analysis for Day 32; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -1551.194, 90% CI 2-sided [-2190.515 to -911.873]
Statistical Analysis 2: Comparison: Placebo vs MEDI0382; Statistical Analysis for Day 59; Test type: Superiority; p = 0.015, ANCOVA; Mean Difference (Net) = -1332.515, 90% CI 2-sided [-2187.711 to -477.318]

4. Secondary Outcome: Percent Change in Total Energy Expenditure (TEE) as Measured by Whole Room Indirect Calorimetry From Baseline to Day 58
Description: A whole room calorimetry assessment was used to measure gaseous exchange while exercising and therefore indirect estimates of energy expenditure over a 24-hour period. For assessment, participants had to enter the whole room calorimeter for up to 36 hours and reside inside for this entire duration (include toilet visits). During the time in the calorimeter participants were asked to exercise on an exercise bike for 15-minute intervals at 4 times. During these sessions participants were asked to aim for a heart rate of 65% of maximum (defined as 220 beats per minute minus age) and complete the full 15-minute session. In addition, participants abstained from caffeinated drinks for at least 24 hours prior to measurements as caffeine may increase energy expenditure (EE) and dietary advice was given to ensure participants had a neutral energy balance prior to whole calorimetry assessments. Percent change in TEE is reported. Day 15 was considered as baseline for this outcome measure.
Time Frame: Baseline (Day 15) and Day 58
Population: mITT population: Participants in the ITT population (who received any study drug) who received at least one dose of the study drug in the double-blind treatment period, and analyzed according to their randomized treatment group. Here, "number of participants analyzed" denotes those participants who were evaluable at baseline and Day 58.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent change in TEE
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 7 | 12
Percent change in TEE | 2.032 [-2.833 to 6.898] | -1.141 [-4.825 to 2.544]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382; Test type: Superiority; p = 0.384, ANCOVA; Mean Difference (Net) = -3.173, 90% CI 2-sided [-9.368 to 3.022]

5. Secondary Outcome: Change in TEE as Measured by Whole Room Indirect Calorimetry From Baseline to Day 58
Description: A whole room calorimetry assessment was used to measure gaseous exchange while exercising and therefore indirect estimates of energy expenditure over a 24-hour period. For the assessment, participants had to enter the whole room calorimeter for up to 36 hours and reside inside for this entire duration (this will include toilet visits too). During the time in the calorimeter participants were asked to exercise on an exercise bike for 15-minute intervals at 4 times. During these sessions participants were asked to aim for a heart rate of 65% of maximum (defined as 220 beats per minute minus age) and complete the full 15-minute session. In addition, participants abstained from caffeinated drinks for at least 24 hours prior to measurements as caffeine may increase EE and dietary advice was given to ensure participants had a neutral energy balance prior to whole calorimetry assessments. Change in TEE is reported. Day 15 was considered as baseline for this outcome measure.
Time Frame: Baseline (Day 15) and Day 58
Population: as for outcome 4
Measure: Least Squares Mean (90% Confidence Interval); unit: kilojoules/kg fat body mass
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 7 | 12
kilojoules/kg fat body mass | 5.969 [-8.364 to 20.302] | -4.070 [-14.924 to 6.783]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382; Test type: Superiority; p = 0.351, ANCOVA; Mean Difference (Net) = -10.039, 90% CI 2-sided [-28.287 to 8.209]

6. Secondary Outcome: Percent Change in Activity Energy Expenditure (AEE) as Measured by Whole Room Indirect Calorimetry From Baseline to Day 58
Description: A whole room calorimetry assessment was used to measure gaseous exchange while exercising and therefore indirect estimates of energy expenditure over a 24-hour period. For the assessment, participants had to enter the whole room calorimeter for up to 36 hours and reside inside for this entire duration (this will include toilet visits too). During the time in the calorimeter participants were asked to exercise on an exercise bike for 15-minute intervals at 4 times. During these sessions participants were asked to aim for a heart rate of 65% of maximum (defined as 220 beats per minute minus age) and complete the full 15-minute session. In addition, participants abstained from caffeinated drinks for at least 24 hours prior to measurements as caffeine may increase EE and dietary advice was given to ensure participants had a neutral energy balance prior to whole calorimetry assessments. Percent change in AEE is reported. Day 15 was considered as baseline for this outcome measure.
Time Frame: Baseline (Day 15) and Day 58
Population: as for outcome 4
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent change in AEE
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 7 | 12
Percent change in AEE | -0.446 [-6.836 to 5.943] | -0.261 [-5.139 to 4.618]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382; Test type: Superiority; p = 0.968, ANCOVA; Mean Difference (Net) = 0.186, 90% CI 2-sided [-7.858 to 8.229]

7. Secondary Outcome: Change in AEE as Measured by Whole Room Indirect Calorimetry From Baseline to Day 58
Description: A whole room calorimetry assessment was used to measure gaseous exchange while exercising and therefore indirect estimates of energy expenditure over a 24-hour period. For the assessment, participants had to enter the whole room calorimeter for up to 36 hours and reside inside for this entire duration (this will include toilet visits too). During the time in the calorimeter participants were asked to exercise on an exercise bike for 15-minute intervals at 4 times. During these sessions participants were asked to aim for a heart rate of 65% of maximum (defined as 220 beats per minute minus age) and complete the full 15-minute session. In addition, participants abstained from caffeinated drinks for at least 24 hours prior to measurements as caffeine may increase EE and dietary advice was given to ensure participants had a neutral energy balance prior to whole calorimetry assessments. Change in AEE is reported. Day 15 was considered as baseline for this outcome measure.
Time Frame: Baseline (Day 15) and Day 58
Population: as for outcome 4
Measure: Least Squares Mean (90% Confidence Interval); unit: kilojoules/kg fat body mass
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 7 | 12
kilojoules/kg fat body mass | -1.132 [-3.259 to 0.995] | -0.265 [-1.889 to 1.359]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382; Test type: Superiority; p = 0.580, ANCOVA; Mean Difference (Net) = 0.867, 90% CI 2-sided [-1.810 to 3.545]

8. Secondary Outcome: Percent Change in Resting Energy Expenditure (REE) as Measured by Whole Room Indirect Calorimetry From Baseline to Day 58
Description: The REE represents the amount of calories required for a 24-hour period by the body during a non-active period and is assessed by whole room indirect calorimetry method. Percent change in REE is reported. Day 15 was considered as baseline for this outcome measure.
Time Frame: Baseline (Day 15) and Day 58
Population: mITT population:Participants in the ITT population (who received any study drug) who received at least one dose of the study drug in the double-blind treatment period, and analyzed according to their randomized treatment group. Here, "number of participants analyzed" denotes those participants who were evaluable at baseline and Day 58.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent change in REE
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 7 | 12
Percent change in REE | 8.113 [3.254 to 12.972] | 4.468 [0.816 to 8.120]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382; Test type: Superiority; p = 0.324, ANCOVA; Mean Difference (Net) = -3.645, 90% CI 2-sided [-9.894 to 2.603]

9. Secondary Outcome: Change in REE as Measured by Whole Room Indirect Calorimetry From Baseline to Day 58
Description: The REE represents the amount of calories required for a 24-hour period by the body during a non-active period and is assessed by whole room indirect calorimetry method. Change in REE is reported. Day 15 was considered as baseline for this outcome measure.
Time Frame: Baseline (Day 15) and Day 58
Population: as for outcome 4
Measure: Least Squares Mean (90% Confidence Interval); unit: kilojoules/kg fat body mass
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 7 | 12
kilojoules/kg fat body mass | 13.237 [4.104 to 22.369] | 7.565 [0.701 to 14.429]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382; Test type: Superiority; p = 0.412, ANCOVA; Mean Difference (Net) = -5.672, 90% CI 2-sided [-17.415 to 6.072]

10. Secondary Outcome: Percent Change in REE as Measured by Hood Indirect Calorimetry From Baseline to Day 32
Description: Hood calorimetry assessment was used to measure REE. A large plastic hood is placed over participants head for 20 minutes and measurements of gaseous exchange are undertaken. Participants were rested for at least 1 hour prior to hood calorimetry measures; during a hood calorimetry assessment the participants were asked to remain quiet and rested for 40 minutes in total with 10 minutes before and after the assessment to allow for room air assessment. Percent change in REE is reported. Day 16 was considered as baseline for this outcome measure.
Time Frame: Baseline (Day 16) and Day 32
Population: mITT population: Participants in the ITT population (who received any study drug) who received at least one dose of the study drug in the double-blind treatment period, and analyzed according to their randomized treatment group. Here, "number of participants analyzed" denotes those participants who were evaluable at baseline and Day 32.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent Change in REE
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 7 | 12
Percent Change in REE | 1.189 [-5.955 to 8.332] | 8.546 [3.138 to 13.954]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382; Test type: Superiority; p = 0.177, ANCOVA; Mean Difference (Net) = 7.357, 90% CI 2-sided [-1.742 to 16.456]

11. Secondary Outcome: Change in REE as Measured by Hood Indirect Calorimetry From Baseline to Day 32
Description: Hood calorimetry assessment was used to measure REE. A large plastic hood is placed over participants head for 20 minutes and measurements of gaseous exchange are undertaken. Participants were rested for at least 1 hour prior to hood calorimetry measures; during a hood calorimetry assessment the participants were asked to remain quiet and rested for 40 minutes in total with 10 minutes before and after the assessment to allow for room air assessment. Change in REE is reported. Day 16 was considered as baseline for this outcome measure.
Time Frame: Baseline (Day 16) and Day 32
Population: as for outcome 10
Measure: Least Squares Mean (90% Confidence Interval); unit: kilojoules/kg fat body mass
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 7 | 12
kilojoules/kg fat body mass | 3.316 [-11.080 to 17.712] | 18.502 [7.604 to 29.400]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382; Test type: Superiority; p = 0.168, ANCOVA; Mean Difference (Net) = 15.186, 90% CI 2-sided [-3.151 to 33.523]

12. Secondary Outcome: Change in Body Weight From Baseline to Day 59
Description: Change in body weight from baseline to Day 59 is reported. Day 17 was considered as baseline for this outcome measure. The LOCF analysis was used for missing data imputation for Day 59.
Time Frame: Baseline (Day 17) and Day 59
Population: mITT population: Participants in the ITT population (who received any study drug) who received at least one dose of the study drug in the double-blind treatment period, and analyzed according to their randomized treatment group. Here, "number of participants analyzed" denotes those participants who were evaluable at baseline and Day 59.
Measure: Least Squares Mean (90% Confidence Interval); unit: kg
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 7 | 14
kg | -1.26 [-2.48 to -0.05] | -3.80 [-4.65 to -2.96]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382; Test type: Superiority; p = 0.009, ANCOVA; Mean Difference (Net) = -2.54, 90% CI 2-sided [-4.05 to -1.03]

13. Secondary Outcome: Percent Change in Total Body Fat Mass as Measured by Dual-energy X-ray Absorptiometry (DXA) From Baseline to Day 59
Description: The total body fat mass was measured in kilograms (kg) using DXA. Participants body was scanned using DXA scanner and total body fat mass was determined. Percent change in total body fat mass is reported. Day -1 was considered as baseline for this outcome measure.
Time Frame: Baseline (Day -1) and Day 59
Population: as for outcome 12
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent change in total body fat mass
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 7 | 12
Percent change in total body fat mass | -4.218 [-8.249 to -0.186] | -9.340 [-12.343 to -6.337]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382; Test type: Superiority; p = 0.107, ANCOVA; Mean Difference (Net) = -5.122, 90% CI 2-sided [-10.364 to 0.119]

14. Secondary Outcome: Change in Total Body Fat Mass as Measured by DXA From Baseline to Day 59
Description: The total body fat mass was measured in kg using DXA. Participants body was scanned using DXA scanner and total body fat mass was determined. Change in total body fat mass is reported. Day -1 was considered as baseline for this outcome measure.
Time Frame: Baseline (Day -1) and Day 59
Population: as for outcome 12
Measure: Least Squares Mean (90% Confidence Interval); unit: Kg
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 7 | 12
Kg | -1.455 [-2.806 to -0.103] | -3.303 [-4.310 to -2.296]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382; Test type: Superiority; p = 0.085, ANCOVA; Mean Difference (Net) = -1.848, 90% CI 2-sided [-3.605 to -0.091]

15. Secondary Outcome: Percent Change in Total Body Fat Mass: Lean Mass Ratio as Measured by DXA From Baseline to Day 59
Description: The total body fat mass and lean body mass was measured in kg using DXA. Participants body was scanned using DXA scanner and total body fat mass and lean mass was determined. Percent change in total body fat mass:lean mass (TBFM:LM) ratio is reported. Day -1 was considered as baseline for this outcome measure.
Time Frame: Baseline (Day -1) and Day 59
Population: as for outcome 12
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent change in TBFM:LM ratio
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 7 | 12
Percent change in TBFM:LM ratio | -1.667 [-4.934 to 1.600] | -4.827 [-7.298 to -2.355]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382; Test type: Superiority; p = 0.204, ANCOVA; Mean Difference (Net) = -3.159, 90% CI 2-sided [-7.326 to 1.007]

16. Secondary Outcome: Change in Total Body Fat Mass: Lean Mass Ratio as Measured by DXA From Baseline to Day 59
Description: The total body fat mass and lean body mass was measured in kg using DXA. Participants body was scanned using DXA scanner and total body fat mass and lean mass was determined. Change in total body fat mass:lean mass (TBFM:LM) ratio is reported. Day -1 was considered as baseline for this outcome measure.
Time Frame: Baseline (Day -1) and Day 59
Population: as for outcome 12
Measure: Least Squares Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 7 | 12
Ratio | -0.010 [-0.027 to 0.007] | -0.029 [-0.042 to -0.016]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382; Test type: Superiority; p = 0.145, ANCOVA; Mean Difference (Net) = -0.019, 90% CI 2-sided [-0.041 to 0.003]

17. Secondary Outcome: Change in Fasting Glucose During a Mixed-meal Tolerance Test (MMTT) From Baseline to Day 59
Description: The MMTT involves consumption of a standardized solid breakfast meal within 5 minutes, following a minimum 12 hours fast, and timed serial blood samples are obtained for measurement of glucose levels through 240 minutes with no additional food intake during this time. Change in fasting glucose is reported. Day -1 was considered as baseline for this outcome measure.
Time Frame: Baseline (Day -1) and Day 59
Population: as for outcome 12
Measure: Least Squares Mean (90% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 7 | 12
mg/dL | -12.600 [-21.673 to -3.527] | -38.601 [-45.360 to -31.842]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382; Test type: Superiority; p = 0.001, ANCOVA; Mean Difference (Net) = -26.001, 90% CI 2-sided [-37.801 to -14.201]

18. Secondary Outcome: Percent Change in Glucose Area Under the Concentration-time Curve at 0 to 4 Hours (AUC0-4hrs) During a MMTT From Baseline to Day 59
Description: The MMTT involves consumption of a standardized solid breakfast meal within 5 minutes, following a minimum 12 hours fast, and timed serial blood samples are obtained for measurement of glucose levels through 240 minutes with no additional food intake during this time. Percent change in glucose AUC0-4hrs during MMTT is reported. Day -1 was considered as baseline for this outcome measure.
Time Frame: Baseline (Day -1) and Day 59
Population: as for outcome 12
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage change in glucose AUC0-4hrs
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 7 | 12
Percentage change in glucose AUC0-4hrs | -6.773 [-12.528 to -1.018] | -19.105 [-23.434 to -14.777]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382; Test type: Superiority; p = 0.010, ANCOVA; Mean Difference (Net) = -12.332, 90% CI 2-sided [-19.726 to -4.938]

19. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life threatening experience immediate risk of dying, persistent or significant disability/incapacity, and congenital anomaly. TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug. From Day 1 to Day 16 all participants in both treatment arms received placebo so that analysis of energy intake in participants who were randomised to MEDI0382 may be performed. Hence, TEAEs were not applicable for Day 1 to Day 16. The TEAEs were recorded and reported for double-blind treatment period ie, from Day 17.
Time Frame: Day 17 through 28 days post last dose (approximately 14 months)
Population: Participants who received any study drug in the double-blind treatment period and were analyzed according to the treatment they received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 7 | 18
Participants
  Any TEAEs | 5 | 17
  Any TESAEs | 0 | 2

20. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs
Description: Number of participants with clinical laboratory abnormalities reported as TEAEs are reported. Clinical laboratory abnormalities are defined as any abnormal findings in analysis of serum chemistry, hematology, and urinalysis. From Day 1 to Day 16 all participants in both treatment arms received placebo so that analysis of energy intake in participants who were randomised to MEDI0382 may be performed. Hence, TEAEs were not applicable for Day 1 to Day 16. The TEAEs were recorded and reported for double-blind treatment period ie, from Day 17.
Time Frame: Day 17 through 28 days post last dose (approximately 14 months)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 7 | 18
Participants | 0 | 0

21. Secondary Outcome: Number of Participants With Abnormal Vital Signs Reported as TEAEs
Description: Number of participants with abnormal vital signs reported as TEAEs are reported. Abnormal vital signs reported as TEAEs included any abnormal findings in body temperature, blood pressure, pulse rate, and respiratory rate. From Day 1 to Day 16 all participants in both treatment arms received placebo so that analysis of energy intake in participants who were randomised to MEDI0382 may be performed. Hence, TEAEs were not applicable for Day 1 to Day 16. The TEAEs were recorded and reported for double-blind treatment period ie, from Day 17.
Time Frame: Day 17 through 28 days post last dose (approximately 14 months)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 7 | 18
Participants | 0 | 0

22. Secondary Outcome: Number of Participants With Abnormal Electrocardiograms (ECGs) Reported as TEAEs
Description: Number of participants with abnormal ECG reported as TEAEs are reported. From Day 1 to Day 16 all participants in both treatment arms received placebo so that analysis of energy intake in participants who were randomised to MEDI0382 may be performed. Hence, TEAEs were not applicable for Day 1 to Day 16. The TEAEs were recorded and reported for double-blind treatment period ie, from Day 17.
Time Frame: Day 17 through 28 days post last dose (approximately 14 months)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 7 | 18
Participants | 0 | 4

23. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADAs) to MEDI0382
Description: Number of participants with positive ADA to MEDI0382 are reported. Treatment-boosted ADA is defined as baseline ADA titer that was boosted to a 4-fold or higher level following drug administration. Treatment-emergent ADA is defined as the sum of treatment-induced ADA (post-baseline positive only) and treatment-boosted ADA. From Day 1 to Day 16 all participants in both treatment arms received placebo so that analysis of energy intake in participants who were randomised to MEDI0382 may be performed. Hence, ADA were not applicable for Day 1 to Day 16. The ADAs were recorded and reported for double-blind treatment period ie, from Day 17.
Time Frame: Day 17 (predose), Day 32 (predose), Day 59; and 28 days post last dose (approximately 14 months)
Population: Participants who received any study drug in the double-blind treatment period and were analyzed according to the treatment they received. Here, "number of participants analyzed" denotes those participants who had post-baseline ADA results.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 7 | 14
Participants
  ADA positive post-BL | 0 | 3
  Treatment-boosted ADA | 0 | 0
  Treatment-emergent ADA | 0 | 3

ADVERSE EVENTS:
Time Frame: Day 17 through 28 days post last dose (approximately 14 months)
Description: From Day 1 to Day 16 all participants in both treatment arms received placebo so that analysis of energy intake in participants who were randomised to MEDI0382 may be performed. Hence, TEAEs were not applicable for Day 1 to Day 16. The TEAEs were recorded and reported for double-blind treatment period ie, from Day 17.
Arm/Group | Placebo | MEDI0382
All-Cause Mortality (participants affected / at risk) | 0/7 | 1/18
Serious Adverse Events (participants affected / at risk) | 0/7 | 2/18
Other Adverse Events (participants affected / at risk) | 5/7 | 16/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=7) | MEDI0382 (N=18)
Coronary artery thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=7) | MEDI0382 (N=18)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Breath odour (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (5)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 3 (6)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Eructation (Gastrointestinal disorders) | 0 (0) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 13 (19)
Retching (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (5)
Injection site erythema (General disorders) | 0 (0) | 2 (2)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (4)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Electrocardiogram t wave amplitude decreased (Investigations) | 0 (0) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (5) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 3 (3)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Coital bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
For Participant Flow section, Pre-assignment details:

Data not collected for Secondary Outcome Measures #24 and #25:

* Percentage change in TEE as measured by doubly labelled water from baseline (Day 17) to End of Treatment (EOT; Day 58 or 59],
* Change in TEE as measured by doubly labelled water from baseline (Day 17) to End of Treatment (EOT; Day 58 or 59]).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises on going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/77/NCT03596177/Prot_002.pdf
  • Statistical Analysis Plan (2019-02-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT03596177/SAP_003.pdf